CLINICAL TRIAL: NCT00183495
Title: Determinants and Manifestation of Illness Behavior in Promoting Treatment Adherence Among Individuals With Bipolar Depression
Brief Title: Understanding Treatment Adherence Among Individuals With Bipolar Disorder
Status: Completed | Type: Observational
Sponsor: Case Western Reserve University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Martha Sajatovic, MD, Professor of Psychiatry, Case Western Reserve University
Other Study IDs: K23MH065599-01 (NIH); K23MH065599-01 (NIH); DAHBR 9K-TA
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Bipolar Disorder
Keywords: Depression, Bipolar; Manic-Depressive Psychosis
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study will examine how various factors, such as psychiatric symptoms, gender, social support, substance use, and attitudes toward medication, affect treatment adherence in individuals with bipolar disorder.

DETAILED DESCRIPTION:
Bipolar Disorder (BPD), also known as manic-depressive illness, is a disorder that causes frequent shifts in an individual's mood, energy, and ability to function. An individual with BPD may go through periods of mania, which are characterized by increased energy, irritability, and an excessively "high" euphoric mood. The manic periods are followed by periods of depression, which are characterized by decreased energy, feelings of hopelessness, and anxiety. BPD is a persistent and severe mental illness with a high suicide rate; it must be strictly managed through medication and therapy. Many BPD medications have been developed recently; however, there are still many individuals who do not respond well to medication treatment. Research has shown that the way individuals experience illness has an effect on their response to medication. The purpose of this study is to gain insight into how individuals with BPD perceive and respond to medication treatment. Factors such as gender, degree of social support, drug and alcohol usage, and attitudes towards medication will be evaluated to understand how they affect medication and treatment adherence.

This 6-month study will consist of 3 interviews. Each interview will last approximately 2 and ½ hours and will include numerous standardized psychological questionnaires. The questionnaires will assess participants' attitudes toward BPD treatment; psychiatric illness severity, including symptoms of mania and depression; level of addiction to alcohol and drugs; availability of social support resources; and medication adherence.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of bipolar disorder type I for at least two years prior to study entry
* Has experienced an index depressive episode
* Received treatment with medication to stabilize mood for at least 6 months prior to study entry
* Able to participate in psychiatric interviews
* Lives in the Northeast Ohio area and is a patient at either Northeast Ohio Health Services or The Mood Disorders Clinic at University Hospitals of Cleveland

Exclusion Criteria:

* Unable/unwilling to participate in psychiatric interviews

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with bipolar disorder receiving treatment at a Community Mental Health Clinic in Northeast Ohio.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2004-03; Primary Completion 2007-03 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Attitudes toward Mood Stabilizers Questionnaire (AMSQ) | Change from Baseline to 6 month visit
  The AMSQ is a 19-item scale which is a modification of the Lithium Attitudes Questionnaire (LAQ) that evaluates an individual's attitude toward mood-stabilizing medication. The questions are in a yes/no format. The AMSQ has 7 subscales that represent key attitudinal domains with respect to adherence, as follows: 1. opposition to prophylaxis, 2. denial of therapeutic effectiveness, 3. fear of adverse effects, 4. difficulty with medication routines, 5. denial of illness severity, 6. negative attitude toward drugs in general, and 7. lack of information about mood stabilizers. Total scores range from 0 to 19. Higher scores on the total and each subscale represent more negative attitudes toward mood stabilizers.
Brief Psychiatric Rating Scale (BPRS) | Change from Baseline to 6 month visit
  The BPRS measures levels of mania. There are 24 items, scored on a 7-point scale ranging from 0 to 6. Total scores range from 0 to 42, with higher scores indicating higher levels of mania.
Addiction Severity Index (ASI) | Change from Baseline to 6 month visit
  A portion of the standardized instrument measuring level of addiction to alcohol and drugs. Items 1-14 of the Alcohol/Drug index were used. The ASI evaluated both lifetime and past-30 day use of a wide variety of commonly abused substances. Each question is divided by its maximum answer value and by the total number of questions in the composite. These individual results are then summed.
  The six questions (A-F) that make up the alcohol composite score is determined by:
  A/180 + B/180 + C/180 + D/24 + E/24 + log F/44.
  The 13 questions (A-M) that make up the drug composite score is determined by:
  A/390 + B/390 + C/390 + D/390 + E/390 + F/390 + G/390 + H/390 + I/390 + J/390 + K/390 + L/52 + M/52.
Interpersonal Suppose Evaluation List (ISEL) | Change from Baseline to 6 month visit
  The ISEL is a 40-item self-report questionnaire that was developed to assess availability of social support resources. A total index is composed of four subscales: tangible assistance (material aid), appraisal (availability of someone to talk to about life's problems), self-esteem (positive appraisal of self from others and positive comparison when comparing one's self with others) and belonging (people with whom one can do things). Response for each item is coded on a 4-point Likert scale ranging from definitely false to definitely true. Total scores range from 0 to 120, with higher scores indicating a higher availability of perceived social support.
Tablets Routine Questionnaire (TRQ) | Change from Baseline to 6 month visit
  The TRQ evaluates adherence to medications via a brief self-report instrument that has been validated in populations with bipolar disorder medication adherence. The TRQ identifies nonadherent individuals, defined as those who miss 30% or more of their medication in the last week or month. Total scores are represented as a percentage and range from 0 to 100, with higher scores indicating a greater level of nonadherence (higher scores indicate worse adherence to medications).
Hamilton Rating Scale for Depression (HAM-D) | Change from Baseline to 6 month visit
  The HAM-D measures form lists 21 items, the scoring is based on the first 17. Eight items are scored on a 5-point scale, ranging from 0 = not present to 4 = severe. Nine are scored from 0-2. Total scores range from 0-52, with higher scores indicating worse depression. The categories are as follows: 0-7 are considered as being normal, 8-16 suggest mild depression, 17-23 moderate depression and scores over 24 are indicative of severe depression; the maximum score is 52.

CONTACTS AND LOCATIONS:
Overall Officials: Martha Sajatovic, MD, Principal Investigator — Case Western Reserve University School of Medicine
Locations (1):
- Northeast Ohio Health Services, Beachwood, Ohio, United States

REFERENCES:
- [Result] Sajatovic M, Ignacio RV, West JA, Cassidy KA, Safavi R, Kilbourne AM, Blow FC. Predictors of nonadherence among individuals with bipolar disorder receiving treatment in a community mental health clinic. Compr Psychiatry. 2009 Mar-Apr;50(2):100-7. doi: 10.1016/j.comppsych.2008.06.008. Epub 2008 Aug 23. PMID 19216885
- [Derived] Smilowitz S, Aftab A, Aebi M, Levin J, Tatsuoka C, Sajatovic M. Age-Related Differences in Medication Adherence, Symptoms, and Stigma in Poorly Adherent Adults With Bipolar Disorder. J Geriatr Psychiatry Neurol. 2020 Sep;33(5):250-255. doi: 10.1177/0891988719874116. Epub 2019 Sep 22. PMID 31542988
- [Derived] Sajatovic M, Tatsuoka C, Cassidy KA, Klein PJ, Fuentes-Casiano E, Cage J, Aebi ME, Ramirez LF, Blixen C, Perzynski AT, Bauer MS, Safren SA, Levin JB. A 6-Month, Prospective, Randomized Controlled Trial of Customized Adherence Enhancement Versus Bipolar-Specific Educational Control in Poorly Adherent Individuals With Bipolar Disorder. J Clin Psychiatry. 2018 Sep 25;79(6):17m12036. doi: 10.4088/JCP.17m12036. PMID 30256551
- [Derived] Sajatovic M, Micula-Gondek W, Tatsuoka C, Bialko C. The relationship of gender and gender identity to treatment adherence among individuals with bipolar disorder. Gend Med. 2011 Aug;8(4):261-8. doi: 10.1016/j.genm.2011.06.002. Epub 2011 Jul 16. PMID 21763217